CLINICAL TRIAL: NCT01022190
Title: Effect of Etoricoxib (Arcoxia) in Preventing Heterotopic Ossification After Total Hip Arthroplasty
Brief Title: Prevention of Heterotopic Ossification With Arcoxia After Total Hip Replacement
Acronym: Arcoxia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Jaap Brunnekreef, PhD, Radboud University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A2009-36182
Record Dates: First submitted 2009-11-27; First posted 2009-12-01 (Estimated); Results first posted 2013-09-02 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Ossification, Heterotopic
Keywords: Arthroplasty; Hip; Cemented; Heterotopic ossification; Selective Cyclooxygenase-2 Inhibitors; Arthroplasty, Replacement; Hip Prosthesis; Cyclooxygenase Inhibitors
MeSH Terms: conditions — Ossification, Heterotopic | interventions — Etoricoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: Etoricoxib (Arcoxia, MSD), 90 mg. (Experimental): Intervention drug: Etoricoxib (Arcoxia, MSD), 90 mg, orally, one time a day, for a 7 day period.
  Interventions: Drug: Etoricoxib (Arcoxia)

INTERVENTIONS:
Drug: Etoricoxib (Arcoxia) — Oral intake of 90 mg Etoricoxib (Arcoxia) during 7-days
  Other Names: Etoricoxib, Arcoxia

SUMMARY:
The purpose of the study is to determine whether Arcoxia is effective in preventing heterotopic ossification after total hip arthroplasty.

DETAILED DESCRIPTION:
Rationale: Heterotopic ossification is a frequent complication after total hip replacement. Nonsteroidal anti-inflammatory drugs (NSAIDs) are known to effectively prevent heterotopic ossification, but gastrointestinal complaints are reported frequently. Selective cyclooxygenase-2 (COX-2) inhibiting NSAID produce less gastrointestinal side effects.

Objective: Preventing heterotopic ossification. Study design: A prospective two-stage study design for phase-2 clinical trials with 42 patients to determine if Arcoxia (a COX-2 inhibitor) 90-mg oral prevents heterotopic ossification. In the first stage, 19-patients are included. Another 23-patients are included when at least 90-percent of patients in first stage have Brooker classification 0, 1 or 2 at 6-months follow-up.

Study population: 42-patients with cemented total hip arthroplasty age 18 - 75 yr old.

Intervention: All subjects receive 90-mg Arcoxia oral for 7-days. Main study parameters/endpoints: The main study parameter is the degree of heterotopic ossification assessed on AP radiographs using the Brooker classification.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: No risks are associated with participating into the research. Besides the oral intake of Arcoxia, no extra burden is associated with participating in the study. The postoperative care does not change. Radiographic examinations will be routinely performed the day before surgery, immediately after operation, at 6-weeks and 6-months after surgery. The degree of heterotopic ossification will be determined by x-ray assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or secondary hip osteoarthritis who are scheduled for cemented total hip replacement at the Radboud University Nijmegen Medical Centre, Nijmegen, the Netherlands.
* Written informed consent is obtained from the patient or the legally accepted representative.

Exclusion Criteria:

* Patients with rheumatoid arthritis, ankylosing spondylitis, or femoral neck fractures
* Patients with previous allergic reaction on non-steroidal anti-inflammatory drugs
* Patients with gastrointestinal complaints at admission, a history of gastrointestinal ulcers or perforations, inflammatory bowel-disease, hepatic dysfunction, renal dysfunction with a clearance below 30 ml/min and cardiac insufficiency.
* Patients with blood pressure consistently > 140/90 mmHg and who have not been adequately controlled.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R.P.H. Veth, Prof, MD, Study Chair — Radboud University Nijmegen Medical Centre, department of Orthopedics
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Background] van der Heide HJ, Rijnberg WJ, Van Sorge A, Van Kampen A, Schreurs BW. Similar effects of rofecoxib and indomethacin on the incidence of heterotopic ossification after hip arthroplasty. Acta Orthop. 2007 Feb;78(1):90-4. doi: 10.1080/17453670610013475. PMID 17453398
- [Background] van der Heide HJ, Koorevaar RC, Lemmens JA, van Kampen A, Schreurs BW. Rofecoxib inhibits heterotopic ossification after total hip arthroplasty. Arch Orthop Trauma Surg. 2007 Sep;127(7):557-61. doi: 10.1007/s00402-006-0243-1. Epub 2006 Nov 16. PMID 17106714
- [Result] Brunnekreef JJ, Hoogervorst P, Ploegmakers MJ, Rijnen WH, Schreurs BW. Is etoricoxib effective in preventing heterotopic ossification after primary total hip arthroplasty? Int Orthop. 2013 Apr;37(4):583-7. doi: 10.1007/s00264-013-1781-0. Epub 2013 Jan 29. PMID 23359100
- See also: Related Info — http://www.umcn.nl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects have been recruited
Pre-assignment Details: No participants were excluded
Groups:
- Etoricoxib, 90 mg, Orally, Ones a Day: Patients who underwent total hip arthroplasty were administered Etoricoxib, 90 mg, orally, one a day for a 7 day period to prevent heterotopic ossification of the hip joint after the operation.
Period: Overall Study
Arm/Group | Etoricoxib, 90 mg, Orally, Ones a Day
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Etoricoxib
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 54.2 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 17
Region of Enrollment [Number; unit: participants]
  Netherlands | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Heterotopic Ossification (HO) at 6 Months Postoperatively.
Description: Percentage of participants in which Heterotopic Ossification of the hip was assessed, according to the Brooker grade.
  Brooker-0): No ossification. Brooker-1): Isolated bone islands, Brooker-2): Bone spurs from the pelvis or proximal femur;space between opposing surface ≥ 1 cm, Brooker-3): Bone spurs from the pelvis or proximal femur;space between opposing surface < 1 cm, Brooker-4): Apparent bony ankylosis. Brooker score 1 to 4 are considered 'heterotopic ossification'.
Time Frame: 6 months postoperatively
Population: Patients who underwent total hip arthroplasty and received afterwards Etoricoxib medication.
Measure: Number; unit: percentage of participants
Groups:
- Etoricoxib, 90 mg, Orally, One a Day for 7 Days Period: Etoricoxib, 90 mg, which was administered orally, for a 7-day period to all participants.
Arm/Group | Etoricoxib, 90 mg, Orally, One a Day for 7 Days Period
Number analyzed (Participants) | 42
percentage of participants | 38

ADVERSE EVENTS:
Arm/Group | Etoricoxib
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

LIMITATIONS AND CAVEATS:
Small sample size. However, due to ethical considerations, a two phase model is necessary to indicate effectivity of Etoricoxib in prevention HO in this phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No